CLINICAL TRIAL: NCT01821898
Title: Eosinophilic Esophagitis Clinical Therapy Comparison Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was below expectation
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carla McGuire Davis, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-27999; 36533 (Other Grant/Funding Number: American Academy of Allergy, Asthama and Immunology)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophil; Reflux; Esophagus; Food allergy; Trouble Swallowing; Pediatrics
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux; Food Hypersensitivity; Deglutition Disorders | interventions — Budesonide; Steroids; Elimination Diets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive for food allergy: Group A (Active Comparator): Oral Budesonide
  Interventions: Drug: Oral Budesonide
- Positive for food allergy: Group B (Active Comparator): Elimination diet
  Interventions: Other: Elimination diet

INTERVENTIONS:
Drug: Oral Budesonide — This group will receive oral viscous budesonide at a dose of 1 or 2 mg depending on the height divided twice a day
  Other Names: Steroid
  Arms: Positive for food allergy: Group A
Other: Elimination diet — This group will receive an elimination diet
  Arms: Positive for food allergy: Group B

SUMMARY:
Eosinophilic Esophagitis (EoE) is a disorder in which a type of white blood cell (eosinophil) involved in allergic reactions, enter and cover the walls of the esophagus (food pipe). As a result, the esophagus becomes swollen and blocked making it difficult to swallow, and this leads to heartburn. In severe cases it can lead to food getting stuck in the esophagus and poor growth or weight loss in children

The main purpose of this research study is to compare the effectiveness of two different types of treatment for EoE:

1. Oral viscous budesonide- which is a steroid medication that has been used to treat asthma. Recently, it has been used as a therapy to treat the eosinophilic inflammation in EoE, and
2. Specific food elimination.

The study will also be looking to see if a blood test is useful in following the progression of EoE. Currently the only way to follow EoE is by repeating endoscopy, which is a more "invasive test."

DETAILED DESCRIPTION:
This study is a open label, randomized, prospective clinical trial comparing the efficacy of a topical steroid preparation to an antigen (food) elimination diet.

A total of 40 participants will be recruited for this study that are positive for food allergens. Study participants will be randomly assigned to treatments as described below, and the duration of each treatment phase will be 16 weeks.

The subjects will be randomized to group A and B. Subject and study team will NOT be blinded to the group assignments.

Group A will receive oral viscous budesonide at a dose of 1 or 2 mg daily depending on the height.

Group B will receive an elimination diet (elimination of the foods the subject is allergic to).

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent and assent if applicable prior to performing any study specific procedure.
2. Male or female subjects aged 3-17 years old.
3. Diagnosis of EoE within 2 months of enrollment (greater than or equal to 15 eosinophils per high powered field in both proximal or distal esophageal specimens).
4. Subjects who have failed at least a two month trial of proton pump inhibitor.
5. A female subject of childbearing potential who is or may become sexually active agrees to routinely use contraception from the time of signing informed consent and assent until 30 days from end of study.
6. Positive allergy testing on prick and/or patch testing.

Exclusion Criteria

1. Subjects who are responsive to at least a two month trial of a proton pump inhibitor.
2. Diagnosis of Inflammatory Bowel Disease or static encephalopathy.
3. Prior abdominal surgery and other organ disorder not including atopic diseases.
4. Previous esophageal surgical procedure.
5. Previous esophageal congenital disorders such as tracheal esophageal fistula and esophageal atresia.
6. Positive for pregnancy.
7. Previous therapy within 6 weeks with oral or swallowed steroids or strict dietary elimination of major allergens
8. Presence of increased eosinophils in the stomach, small intestine, large intestine, and colon based on Debrosse et al.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla M. Davis, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive for Food Allergy: Group A: Oral Budesonide
  Oral Budesonide: This group will receive oral viscous budesonide at a dose of 1 or 2 mg depending on the height divided twice a day. Children < 10 years will receive 1 mg daily. Children 10 years and older will receive 2 mg daily.
Period: Overall Study
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
EoE endoscopy score [Number; unit: cells/high powered field] — The range is 0-300 eosinophils per high powered field and higher numbers correlate with worse outcome. A diagnosis of EoE by endoscopic biopsy is demonstrated by intraepithelial eosinophilic infiltration (peak cell count ≥15 eosinophils/high power field [eos/hpf]).
  cells/high powered field
    Patient 1 | 18 | 0 | 18
    Patient 2 | 0 | 21 | 21
    Patient 3 | 30 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Peak Number of Eosinophils/High Powered Field
Description: The primary outcome will be the peak eosinophil/high powered field on repeat biopsy after the treatment phase.
Time Frame: 16 weeks
Population: None of the enrolled participants had a repeat biopsy because they did not finish the trial due to undue stress and anxiety.
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life Survey Score
Description: PedsQL total survey score to assess overall quality of life before and after treatment
Time Frame: 16 weeks
Population: None of the enrolled participants had a PedQL because they did not finish the trial due to undue stress and anxiety.
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Symptom Score
Description: Assess the subject's symptoms using the validated tool termed Pediatric Eosinophilic Esophagitis (EoE) Symptom Severity Module by measuring % of normal bolus transit swallow and % of normal peristaltic esophageal body contractions.
Time Frame: 16 weeks
Population: Pediatric Eosinophilic Esophagitis (EoE) Symptom Severity Module was not completed because the subjects did not finish the trial due to undue stress and anxiety.
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Exploratory Studies
Description: Proteomic studies search for certain proteins in the blood that may be linked to active EoE. Immune analysis will help identify better methods for diagnosis, treatment, and prevention of immune system changes leading to diseases.
Time Frame: Conclusion of study
Population: Analysis was not performed.
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not collected due to the termination of the study.
Description: Adverse events were not collected due to the termination of the study.
Arm/Group | Positive for Food Allergy: Group A | Positive for Food Allergy: Group B
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial was terminated due to the inability of current subjects to complete the protocol and poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT01821898/Prot_SAP_000.pdf